CLINICAL TRIAL: NCT06392776
Title: Early Diagnosis and Treatment of Undiagnosed Asthma or COPD: THE UCAP 2 TRIAL
Acronym: UCAP2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Protocol ID 4373
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early diagnosis of previously undiagnosed asthma or COPD (Experimental): On the day of randomization the participant will receive a copy of their interpreted spirometry report with a listed diagnosis. This report will be sent to their primary-care practitioner. In addition to the spirometry interpretation, the primary-care practitioner will be provided with a brief one-page guideline-based tool providing advice for pharmacologic and non-pharmacologic treatment of newly diagnosed asthma or COPD. The primary-care practitioner will be encouraged to see the participant as soon as possible to provide care. The participant will similarly be encouraged to make an appointment with the primary-care practitioner as soon as possible to access care for their condition
  Interventions: Other: Early diagnosis and treatment
- Delayed diagnosis of previously undiagnosed asthma or COPD (No Intervention): At the 12 week visit, participants randomized to the delayed diagnosis will complete the trial outcome assessments. After completing the 12 week final trial assessments they will be seen by the study respirologist and treated for their newly diagnosed asthma or COPD.

INTERVENTIONS:
Other: Early diagnosis and treatment — Early diagnosis of previously undiagnosed asthma or COPD and subsequent treatment by a primary care practitioner
  Arms: Early diagnosis of previously undiagnosed asthma or COPD

SUMMARY:
Our research group has found that Canadians with undiagnosed asthma or chronic obstructive pulmonary disease (COPD) have increased respiratory symptoms and worse health-related quality of life.

The investigators recently developed and validated an on-line questionnaire to accurately identify these symptomatic, undiagnosed individuals.

The investigators will advertise in the community asking individuals to complete the on-line questionnaire at home, at their leisure, to determine if they are at risk of asthma or COPD. Those at risk will be invited to participate in a randomized, controlled clinical trial to determine whether early diagnosis of previously undiagnosed asthma or COPD and subsequent treatment by the primary care practitioner will improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years old
* Individuals must be symptomatic with respiratory symptoms
* Individuals must complete the UCAP-Q questionnaire and score a ≥ 6% probability of having either asthma or COPD.
* Individuals who have given written informed consent to participate in this trial in accordance with local regulations;
* Individual must be able to perform pre and post bronchodilator spirometry to measure lung function

Additional Inclusion Criteria for the Randomized Controlled Trial (RCT):

* Individuals who have undiagnosed airflow obstruction on spirometry testing (i.e. Asthma or COPD) will be asked to participate in the RCT.

Exclusion Criteria:

* Individuals who report a previous diagnosis of asthma, COPD, history of lung cancer, bronchiectasis, interstitial lung disease, cystic fibrosis or other significant diagnosed lung disease.
* Individuals currently under the care of a Respirologist.
* Individuals currently using inhaled corticosteroids or long-acting bronchodilators.
* Individuals with history of myocardial infarction, stroke, aortic or cerebral aneurysm, or detached retina or eye surgery within the past 3 months (spirometry is contraindicated)
* Individuals who are in the third trimester of pregnancy
* Individuals involved in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in disease-specific quality of life quantified using the St. George's Respiratory Questionnaire (SGRQ). | 12 weeks
  The change in disease-specific quality of life will be expressed as the total St. George's Respiratory Questionnaire score at 12 weeks minus the score on the day of randomization. This questionnaire includes 3 domains: symptoms (distress caused by specific respiratory symptoms); activity (physical activities that cause or are limited by breathlessness); and impact (social and psychological effects of the respiratory disease). A total change of - 4 points in the SGRQ total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate poor health status.

SECONDARY OUTCOMES:
Changes in overall respiratory symptoms (including cough, sputum and dyspnea) will be assessed using the COPD Assessment Test (CAT) | 12 weeks
  The change in overall respiratory symptom burden will be expressed as the total score of the COPD Assessment Test at 12 weeks minus the score on the day of randomization. A total change of - 2 points in the CAT total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate higher burden.
Changes in forced expiratory volume in one second (FEV1) measured in litres (L) using pre bronchodilator spirometry testing and post bronchodilator spirometry testing. | 12 weeks
  The change will be expressed as the mean change in the FEV1 measurements at 12 weeks in comparison to the lung function measurements on the day of randomization.
Differences between the experimental group and the control group in patient-initiated urgent healthcare utilization events for respiratory illness over the 12-week trial period. | 12 weeks
  Differences between groups in patient-initiated urgent healthcare utilization events for respiratory illness over the 12-week trial period.
Change in dyspnea as assessed by The Baseline and Transitional Dyspnea Indexes | 12 weeks
  The baseline dyspnea index (BDI) is used to rate the severity of dyspnea at a single point in time and the transitional dyspnea index (TDI) is used to assess change in dyspnea at 12 weeks.
  The differences between the experimental group and the control group TDI measured at 12 weeks.
Changes in absenteeism and presenteeism as assessed by the Work Productivity and Activity Impairment Questionnaire (WPAI) | 12 weeks
  The change in absenteeism and presenteeism will be assessed over the 12 week study period. Higher scores indicate greater impairment in work productivity and daily activities
Quality of life changes as assessed by the 36-Item Short Form Health Survey (SF-36) Health Survey Questionnaire | 12 weeks
  The change in general health status will be expressed as the total score of the SF-36 Health Survey Questionnaire at 12 weeks minus the score on the day of randomization. A total change of 8-10 points in the SF-36 has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Aaron, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (4):
- Canada (4):
  - St. Joseph's Hamilton Healthcare, Hamilton, Ontario
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec